CLINICAL TRIAL: NCT06637059
Title: Construction of an Artificially Intelligent Model for Accurate Detection of HCC by Integrating Clinical, Radiological, and Peripheral Immunological Features
Brief Title: Artificially Intelligent Model for Accurate Detection of HCC
Status: Completed | Type: Observational
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, TingBo Liang, Professor, Zhejiang University
Other Study IDs: MMFAIHCC
Record Dates: First submitted 2024-10-05; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: Hepatocellular carcinoma; Early detection; Multi-modal; Fusion model; Artificial intelligence
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Training cohort
  Interventions: Other: observational study
- Internal validation cohort
  Interventions: Other: observational study
- External validation cohort
  Interventions: Other: observational study

INTERVENTIONS:
Other: observational study — observation alone

SUMMARY:
Purpose: Integrating comprehensive information on hepatocellular carcinoma (HCC) is essential to improve its early detection. The investigators aimed to develop a model with multi-modal features (MMF) using artificial intelligence (AI) approaches to enhance the performance of HCC detection.

Experimental Design: A total of 1,092 participants were enrolled from 16 centers. These participants were allocated into the training, internal validation, and external validation cohorts. Peripheral blood specimens were collected prospectively and subjected to mass cytometry analysis. Clinical and radiological data were obtained from electrical medical records. Various AI methods were employed to identify pertinent features and construct single-modal models with optimal performance. The XGBoost algorithm was utilized to amalgamate these models, integrating multi-modal information and facilitating the development of a fusion model. Model evaluation and interpretability were demonstrated using the SHapley Additive exPlanations method.

ELIGIBILITY:
Inclusion Criteria:

* Benign liver diseases, including but not limited to, hemangiomas, hepatic cysts, focal nodular hyperplasia, and cirrhosis

Exclusion Criteria:

* Participants who had undergone previous treatment for HCC or benign liver diseases,
* had taken medications affecting the hematological system within 2 weeks
* those who had received a blood transfusion within 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Benign liver diseases, including but not limited to, hemangiomas, hepatic cysts, focal nodular hyperplasia, and cirrhosis were considered in this study. Participants who had undergone previous treatment for HCC or benign liver diseases, those who had taken medications affecting the hematological system within 2 weeks, or those who had received a blood transfusion within 6 months were excluded from the study.
Sampling Method: Non-Probability Sample
Enrollment: 1092 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Diagnosis of liver disease through CT imaging | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No